CLINICAL TRIAL: NCT00406601
Title: Phase II Prospective Study With BAY-43-9006 in Advanced, Metastatic Soft Tissue Sarcomas, After Anthracycline-based Therapy
Brief Title: BAY-43-9006 in Advanced, Metastatic Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2006-002; EUDRACT 2006-004437-15
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sorafenib (BAY-43-9006) — 800 mg/die orally on a continuous basis

SUMMARY:
The aim of this study (*) is to evaluate the progression free survival rate at 6 months, response rate, overall disease control rate, overall survival of BAY-43-9006 in soft tissue sarcoma patients.

(*) as per Protocol Amendment No. 1 of 16 April 2007 approved by local IEC on 24 July 2007

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, progressive, advanced or metastatic sarcoma after adjuvant and/or first line anthracycline-based regimen; age >=18 yrs; ECOG PS =2; at least 1 measurable target lesion; life expectancy >=12 wks; adequate medullary liver and renal function; written informed consent.

Exclusion Criteria:

* metastatic brain disease; pregnant or breast-feeding patients; serious infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate | at 6 months after enrollment

SECONDARY OUTCOMES:
Overall response rate, overall disease control rate, overall survival | Tumor assessment, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Antman KH. Adjuvant therapy of sarcomas of soft tissue. Semin Oncol. 1997 Oct;24(5):556-60. PMID 9344322
- [Background] Santoro A, Tursz T, Mouridsen H, Verweij J, Steward W, Somers R, Buesa J, Casali P, Spooner D, Rankin E, et al. Doxorubicin versus CYVADIC versus doxorubicin plus ifosfamide in first-line treatment of advanced soft tissue sarcomas: a randomized study of the European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 1995 Jul;13(7):1537-45. doi: 10.1200/JCO.1995.13.7.1537. PMID 7602342